CLINICAL TRIAL: NCT02380768
Title: A Randomized Comparison of the Ambu AuraGain™ and LMA Supreme™ in Infants and Children
Brief Title: A Comparison of the Ambu AuraGain Versus LMA Supreme in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Narasimhan Jagannathan, Primary Investigator; M.D., Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IRB 2015-252
Record Dates: First submitted 2015-02-26; First posted 2015-03-05 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-07

CONDITIONS: Supraglottic Airway
Keywords: Supraglottic airway; Laryngeal mask airway; Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ambu AuraGain (Experimental): Subjects will receive the Ambu AuraGain size 1.5 or 2.0 based on manufacturer guidelines
  Interventions: Device: Ambu AuraGain (size 1.5 or size 2.0)
- LMA Supreme (Active Comparator): Subjects will receive the Ambu AuraGain size 1.5 or 2.0 based on manufacturer guidelines
  Interventions: Device: LMA Supreme (size 1.5 or size 2.0)

INTERVENTIONS:
Device: Ambu AuraGain (size 1.5 or size 2.0) — The device will be inserted and timed. A leak pressure test will be performed after successful insertion and after 10 minutes. The larynx will be visualized by placing a fiberoptic bronchoscope through the device. A gastric tube will be inserted through the device and timed.
  Other Names: Ambu AuraGain
  Arms: Ambu AuraGain
Device: LMA Supreme (size 1.5 or size 2.0) — The device will be inserted and timed. A leak pressure test will be performed after successful insertion and after 10 minutes. The larynx will be visualized by placing a fiberoptic bronchoscope through the device. A gastric tube will be inserted through the device and timed.
  Other Names: LMA Supreme
  Arms: LMA Supreme

SUMMARY:
The purpose of this study is to determine whether there is a clinically relevant difference in airway leak pressures between the Ambu AuraGain and the Laryngeal Mask Airway (LMA) Supreme.

DETAILED DESCRIPTION:
The goal of this prospective randomized study is to compare whether there is a clinically relevant difference in airway leak pressures between the Ambu AuraGain (sizes 1.5 and 2) and the Laryngeal Mask Airway (LMA) Supreme. Parameters of clinical relevance such as insertion success rates, fiberoptic view of the glottic opening, ease and speed of gastric tube placement, airway stability, and peri-operative complications will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for surgery utilizing a supraglottic airway device
* ASA (American Society of Anesthesiologists) I-III classification
* Weighing between 5 - 20 kilograms

Exclusion Criteria:

* Active respiratory infection
* History of difficult mask ventilation
* Diagnosis of congenital syndrome with difficult airway management
* Active gastrointestinal reflux
* Coagulopathy
* Significant Pulmonary disease
* Emergent surgery

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal (airway) leak pressure - Initial | Assessed intraoperatively at the time of confirmed device placement
  The airway pressure at which an airway leak is observed after successful placement of the supraglottic airway
Oropharyngeal (airway) leak pressure - 10 Minutes | Assessed intraoperatively, 10 minutes after the initial confirmed placement of the device
  The airway pressure at which an airway leak is observed 10 minutes after successful placement of the supraglottic airway

SECONDARY OUTCOMES:
Time for Successful Placement of the Supraglottic Airway | Assessed intraoperatively at the time of confirmed device placement
  Time for successful placement of supraglottic device will be recorded
Number of attempts to placement of Supraglottic Airway | Assessed intraoperatively at the time of confirmed device placement
  Number of attempts and insertion techniques will be recorded (maximum of 3 attempts)
Fiberoptic Grade of Laryngeal View through Supraglottic Airway | Assessed intraoperatively at the time of confirmed device placement
  Fiberoptic Grade of Laryngeal View through either device will be graded using a previously published grading system
Gastric Tube Insertion Ease of Placement | Assessed intraoperatively at the time of confirmed gastric tube placement
  The ease of placement, based on a 1-4 scale, will be recorded following placement and confirmation of the gastric tube.
Gastric Tube Insertion Time | Assessed intraoperatively at the time of confirmed gastric tube placement
  The elapsed time from beginning insertion of the gastric tube to confirmation, will be recorded. Confirmation of gastric tube placement will be determined by injection of air with auscultation (listening for sounds) over the stomach with a stethoscope.
Gastric Tube Insertion Attempts | Assessed intraoperatively at the time of confirmed gastric tube placement
  Number of insertion attempts of the gastric tube through the SGA will be recorded. Confirmation of gastric tube placement will be determined by injection of air with auscultation (listening for sounds) over the stomach with a stethoscope.
Postoperative Complications | Participants will be followed for the duration of hospital stay. Outcome measure will be assessed postoperatively in recovery unit.
  Patient will be evaluated for sore throat, cough, dysphonia, stridor, or other airway related complications during the post-operative period.
Intraoperative Complications | Assessed intraoperatively
  Complications such as reflex activation of the airway (coughing, breath holding, laryngospasm, bronchospasm), oxygen desaturation will be recorded, if they occur.

CONTACTS AND LOCATIONS:
Overall Officials: Narasimhan Jagannathan, M.D., Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] White MC, Cook TM, Stoddart PA. A critique of elective pediatric supraglottic airway devices. Paediatr Anaesth. 2009 Jul;19 Suppl 1:55-65. doi: 10.1111/j.1460-9592.2009.02997.x. PMID 19572845
- [Background] Jagannathan N, Ramsey MA, White MC, Sohn L. An update on newer pediatric supraglottic airways with recommendations for clinical use. Paediatr Anaesth. 2015 Apr;25(4):334-45. doi: 10.1111/pan.12614. Epub 2015 Jan 13. PMID 25585975
- [Background] Jagannathan N, Sohn LE, Sawardekar A, Gordon J, Langen KE, Anderson K. A randomised comparison of the LMA SupremeTM and LMAProSealTM in children. Anaesthesia. 2012 Jun;67(6):632-9. doi: 10.1111/j.1365-2044.2012.07088.x. Epub 2012 Mar 15. PMID 22420717
- [Background] Jagannathan N, Sohn L, Sommers K, Belvis D, Shah RD, Sawardekar A, Eidem J, Dagraca J, Mukherji I. A randomized comparison of the laryngeal mask airway supreme and laryngeal mask airway unique in infants and children: does cuff pressure influence leak pressure? Paediatr Anaesth. 2013 Oct;23(10):927-33. doi: 10.1111/pan.12145. Epub 2013 Mar 23. PMID 23521105